CLINICAL TRIAL: NCT04352361
Title: A Single-dose Study to Investigate the Tolerance and Pharmacokinetics of TVB-2640 Tablets in Chinese Healthy Subjects
Brief Title: Ascending Single-dose Study to Evaluate TVB-2640 in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3V2640-CLIN-005-（I）-PK
Record Dates: First submitted 2020-04-14; First posted 2020-04-20 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-04

CONDITIONS: Healthy
MeSH Terms: interventions — TVB-2640

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TVB-2640 tablets (Experimental)
  Interventions: Drug: TVB-2640
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TVB-2640 — TVB-2640 tablets (25mg/50mg/75mg) one tablet at a time, once per day.
  Arms: TVB-2640 tablets
Drug: Placebo — Oral, matching number of placebo Tablets with active arm.
  Arms: placebo

SUMMARY:
Ascending oral single-dose study to evaluate the safety and pharmacokinetics of TVB- 2640 tablets in the Chinese healthy population.

DETAILED DESCRIPTION:
This study is designed as a single-center, randomized, single-blind, placebo-controlled, single-dose escalation trial. The dose groups are 25 mg, 50 mg and 75 mg respectively. The next dose should be tested only if the previous dose has demonstrated to be safe and tolerated, and each subject will receive either the experimental drug or a placebo only once.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 45 (including 18 and 45), both male and female(The 50mg dose half male and half female).
2. Male weight ≥50 kg, female weight ≥45 kg; BMI between 19 and 24 kg/m2 (including boundary value).
3. Those who have no family planning within half a year and are willing to take effective contraceptive measures within half a year after the last administration.
4. Non-pregnant or lactating women.
5. Voluntarily signing the informed consent.

Exclusion Criteria:

1. Persons who have or are currently suffering from any serious clinical diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry and metabolic abnormalities or any other diseases (eye diseases such as corneal edema, keratitis, uveitis etc.) that can interfere with the test results.
2. Previous corneal surgery, gastrointestinal surgery, vagus neurotomy, intestinal resection or any surgical operation that may interfere with gastrointestinal peristalsis, pH or absorption (except hernia repair, appendectomy).
3. Persons with allergic constitution, including those with allergic history of drugs, food or other substances.
4. Those who have used any prescription drugs, over-the-counter drugs, any vitamin products or herbs within 14 days prior to administration.
5. Any drugs that inhibit or induce the liver to metabolize drugs (e.g., inducers - barbiturates, carbamazepine, phenytoin sodium, rifampicin) were used within 30 days prior to administration; Inhibitors - SSRI antidepressants, cimetidine, cyclosporine, macrolides, verapamil, quinolones, pyrrole antifungal agents, HIV protease inhibitors, etc.), p-gp inducers (including rifampicin, st. John's wort, okazepine, and modafinil).
6. Smokers or those who smoked more than 5 cigarettes per day in the 3 months before the study.
7. Alcoholics or regular drinkers in the 6 months prior to the trial, i.e., drinking more than 14 units of alcohol per week (1 unit =360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine).
8. Drinking excessive amounts of tea, coffee or caffeinated beverages (more than 8 cups, 1 cup =250 mL) every day for 3 months before the first administration.
9. Anyone who has consumed or plans to consume any food or beverage containing caffeine (such as coffee, strong tea, chocolate, etc.) or foods rich in xanthine (such as sardines, animal livers, etc.) or beverages within 48 hours prior to the first use of the study drug.
10. Had consumed or planned to consume grapefruit or grapefruit-related citrus fruits (such as lime, grapefruit), star fruit, papaya, pomegranate or more fruit products within 3 days prior to administration.
11. Patients who had donated blood or lost more than 400ml of blood within 3 months before administration.
12. Patients who had participated in other clinical trials and received the study drug treatment within 3 months prior to the initial administration.
13. Those who had used the first oral contraceptive pill within 30 days prior to the first administration, or those who had used long-acting estrogen or progesterone injections or implants within 6 months prior to the first administration.
14. Those who had unprotected sex within 14 days before the first administration (female).
15. Those who have special requirements on diet and cannot follow the unified diet.
16. Those who have worn contact lenses or contact lenses within 7 days before medication administration.
17. Those who fail the alcohol test or abuse the positive drug screening.
18. Abnormal vital signs with clinical significance (normal range: 90 mmHg≤ systolic blood pressure <140 mmHg, 60 mmHg≤ diastolic blood pressure <90 mmHg, 60 beats/min ≤ pulse (resting) ≤100 beats/min;(subject to the judgment of the study physician) or medical examination, electrocardiogram, laboratory examination, breathalyzer test, drug abuse screening, etc.
19. In addition to the above, the researchers judged that the patients were not suitable to participate in the clinical trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 50mg dose: half male and half female.
Enrollment: 34 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and tolerability of TVB-2640 in Chinese healthy volunteers: adverse events and serious adverse events | Up to 4 days
  Evaluation of number of patients reported with adverse events and serious adverse events.

SECONDARY OUTCOMES:
Evaluate the Cmax of TVB-2640 | Up to 3 days
  Evaluate the Peak Plasma Concentration after a single oral dose of TVB-2640 administered to Chinese healthy volunteers.
Tmax of TVB-2640 | Up to 3 days
  Evaluate the Time to reach the maximum plasma concentration after a single oral dose of TVB-2640 administered to Chinese healthy volunteers.
AUC of TVB-2640 | Up to 3 days
  Evaluate the Area under the plasma concentration versus time curve after a single oral dose of TVB-2640 administered to Chinese healthy volunteers.
t1/2 of TVB-2640 | Up to 3 days
  Evaluate the Terminal-Phase Half-Life after a single oral dose of TVB-2640 administered to Chinese healthy volunteers.
CL/F of TVB-2640 | Up to 3 days
  Evaluate the Apparent Systemic Clearance after a single oral dose of TVB-2640 administered to Chinese healthy volunteers.
Vd/F of TVB-2640 | Up to 3 days
  Evaluate the Apparent Volume of Distribution after a single oral dose of TVB-2640 administered to Chinese healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Yahong Chen, MD, Study Director — Ascletis Pharmaceuticals Co., Ltd.
Locations (1):
- Hunan provincial people's hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided